CLINICAL TRIAL: NCT06660563
Title: A Phase 1b Study of JNJ-80948543 in Combination With Other CD3 T-Cell Engagers (TCEs) in Participants With Relapsed/Refractory B-Cell Non-Hodgkin Lymphoid (R/R B-Cell NHL) Malignancies
Brief Title: A Study of JNJ-80948543 in Combination With Other CD3 T-Cell Engagers in Participants With Relapsed/Refractory B-Cell Non-Hodgkin Lymphoma (R/R B-Cell NHL)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 80948543LYM1002; 80948543LYM1002 (Other: Janssen Research & Development, LLC); 2024-514176-41-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma, Non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- JNJ-80948543 (Experimental): Participants will receive JNJ-80948543 in combination with JNJ-75348780 to determine the recommended phase 2 regimen (RP2R) in Part 1 (Dose escalation). JNJ-80948543 will be dosed in an escalation manner in combination with fixed doses of JNJ-75348780. In Part 2 (Dose expansion) participants will receive RP2R of JNJ-80948543 as determined in Part 1 in combination with JNJ-75348780.
  Interventions: Drug: JNJ-80948543; Drug: JNJ-75348780

INTERVENTIONS:
Drug: JNJ-80948543 — JNJ-80948543 will be administered as subcutaneous (SC) or intravenous (IV) injection.
Drug: JNJ-75348780 — JNJ-75348780 will be administered as SC injection.

SUMMARY:
The purpose of this study is to determine the recommended phase 2 regimen (RP2R) for JNJ-80948543 in combination with JNJ-75348780 (Part 1: Dose Escalation) and to further assess the safety of JNJ-80948543 at the RP2R in combination with JNJ-75348780 (Part 2: Dose Expansion).

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of diffuse large B-cell lymphoma (DLBCL), including high-grade B-cell lymphoma and DLBCL arising from indolent lymphoma. All participants must have received at least 2 prior lines of therapy
* Participants must have measurable disease as defined by the appropriate disease response criteria
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Hematologic laboratory parameters must meet the required criterias and the values must be without a transfusion or growth factors for at least 7 days prior to the first dose of study drug
* Participants of childbearing potential must have a negative highly sensitive serum pregnancy test (beta (β)-human chorionic gonadotropin) at screening and within 24 hours before the first dose of study treatment and must agree to further serum or urine pregnancy tests during the study

Exclusion Criteria:

* Known active central nervous system involvement (CNS) or leptomeningeal involvement
* Prior solid-organ transplantation
* Autoimmune or inflammatory disease requiring systemic steroids or other immunosuppressive agents (example, methotrexate or tacrolimus) within 1 year prior to first dose of study drug
* Toxicity from prior anticancer therapy has not resolved to baseline levels or to Grade <= 1 (except alopecia, vitiligo, peripheral neuropathy, or endocrinopathies that are stable on hormone replacement, which may be Grade 2)
* Clinically significant pulmonary compromise defined as the need for supplemental oxygen to maintain adequate oxygenation
* Evidence of clinically significant and/or symptomatic infection (viral, bacterial, or fungal) at the time of study drug initiation. Anti-microbial treatment for infection must be discontinued at least 7 days before the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-01-19 (Estimated); Study Completion 2026-09-21 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicity (DLT) | Up to 1 year and 10 months
  Number of participants with DLT will be reported. DLTs are defined as any of the treatment-related toxicities: any toxicity that would require discontinuation of treatment; Fatal toxicity; Non-hematologic toxicity (Grade 3 toxicity or higher with exceptions); and Hematologic Toxicity (Grade 4 neutrophil count decrease; Grade 4 febrile neutropenia; Grade 3 febrile neutropenia that does not recover with best supportive care within 7 days; Grade 4 platelet count decrease for >=7 days or Grade >3 with Grade >=2 bleeding; Grade 4 anemia).
Number of Participants with Adverse Events (AEs) | Up to 1 year and 10 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.

SECONDARY OUTCOMES:
Serum Concentration of JNJ-80948543 and JNJ-75348780 | Up to 1 year and 10 months
  Serum Concentration for JNJ-80948543 and JNJ-75348780 will be reported.
Area Under the Curve (AUCtau) for JNJ-80948543 and JNJ-75348780 | Up to 1 year and 10 months
  AUC tau is defined as area under the serum concentration-time curve during a dosing interval for JNJ-80948543 and JNJ-75348780.
Maximum Serum Concentration (Cmax) for JNJ-80948543 and JNJ-75348780 | Up to 1 year and 10 months
  Cmax for JNJ-80948543 and JNJ-75348780 will be reported.
Time to Reach Cmax (Tmax) for JNJ-80948543 and JNJ-75348780 | Up to 1 year and 10 months
  Tmax is the time to reach maximum observed serum concentration for JNJ-80948543 and JNJ-75348780.
Number of Participants with Presence of Anti-Drug Antibodies of JNJ-80948543 and JNJ-75348780 | Up to 1 year and 10 months
  Number of participants with presence of anti-drug antibodies of JNJ-80948543 and JNJ-75348780 will be assessed.
Overall Response Rate (ORR) | Up to 1 year and 10 months
  ORR is defined as the percentage of participants who have a best response of partial response (PR) or better as assessed by the investigator based on standard response criteria.
Complete Response Rate (CRR) | Up to 1 year and 10 months
  CR is defined as the percentage of participants who achieve a best response of CR as assessed by the investigator based on standard response criteria.
Duration of Response (DoR) | Up to 1 year and 10 months
  DOR is defined as the time from the first efficacy evaluation at which the participant meet all criteria for a response of PR or better to the date of first documented evidence of progressive disease or death as assessed by the investigator based on standard response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (11):
- Australia (3):
  - Concord Hospital, Concord
  - St Vincents Hospital Melbourne, Fitzroy
  - Macquarie University Hospital, North Ryde
- Spain (5):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Clinic de Barcelona, Barcelona
  - Inst. Cat. Doncologia-H Duran I Reynals, L'Hospitalet de Llobregat
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- University Hospitals Of Leicester Nhs Trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency